CLINICAL TRIAL: NCT02341092
Title: AVEC-TC : Post-traumatic Behavioral Disorders : Analysis and Valuation of the Expertise of Use of the Close Relations of People Victims of Traumatic Brain Injury
Brief Title: Analysis and Valuation of the Expertise of Use of the Close Friends of People Victims of Traumatic Brain Injury
Acronym: AVEC-TC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2012/34
Record Dates: First submitted 2015-01-08; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Traumatic brain injury — Collection of the use of expertise relatives of victims of traumatic brain injury

SUMMARY:
Post-traumatic behavioral disorders : analysis and valuation of the expertise of use of the close friends of people victims of traumatic brain injury.

DETAILED DESCRIPTION:
Collection of the expertise of use of the close friends of people victims of traumatic brain injury. The objective of the work is to collect, to describe, to analyze the corpus of knowledge of the close friends and to transcribe it in two registers, theoretical and practical..

ELIGIBILITY:
Inclusion Criteria:

* Victim of a grave or moderate traumatic brain injury.
* Living at home or in institution
* Seen in consultation in the UH of Angers in neurology and/or in the center of rehabilitation specialized the Capuins and/or followed by Arch Anjou and/or sent by the associations of families.
* 18 - 65 years at the time of the inclusion
* Moderate or grave traumatic brain injury, defined by the score of initial Glasgow 13 and/or a hospitalization of at least 48 hours in intensive care.
* Existence of at least a referent Close friend(relation) : parent(relative), child, spouse, professionnal or other.
* Obtaining of the informed consent of the cranial traumatized, the close friend and the guardian if necessary.

Exclusion Criteria:

* Lack of consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Victim of a grave or moderate traumatic brain injury and existence of at least a referent close friend (relation): parent (relative), child, spouse, professionnal, other.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Collection of the expertise of the close friends(relations) of people victims of a post traumatic brain injury. | 1 day
  The main assessment criteria will be the definition of a list of skills to acquire on behalf of close friends(relations) of a person with a post traumatic brain injury to face, warn and adapt itself to the behavior disorders pos traumatic.

SECONDARY OUTCOMES:
Evaluation of the adequacy of therapeutic medicinal with the recommendations . | 1 Day
  Assessment criteria for the evaluation of the use of the therapeutic and their adequacy with the recommendations will be:
  * Patients percentage under psychotropics
  * Patients percentage under neuroleptic first generation
Evaluation of the resounding of the disorders(confusions) on the social participation. | 1 Day
  Assessment criteria for the resounding of the disorders(confusions) on the social participation will be:
  * The scores Qolibri
  * The scores CIQ
  * The correlation between scores ISDC and Qolibri
  * The correlation between score ISDC and the SF36 score of quality of life of the close friends(relations)
  * The correlation between score ISDC and CIQ
Quantification of the frequency of the post-traumatic behavior disorders. | One day
  The assessment criteria for the quantification of the frequency of the behavior disorders will be the ISDC score (Inventory of dysexecutive syndrome).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Richard-Crémieux, Md-PHD, Principal Investigator — University Hospital, Angers
Locations (1):
- Les Capucins, Angers, Pays de la Loire Region, France

REFERENCES:
- [Result] Saout V, Gambart G, Leguay D, Ferrapie AL, Launay C, Richard I. Aggressive behavior after traumatic brain injury. Ann Phys Rehabil Med. 2011 Jun;54(4):259-69. doi: 10.1016/j.rehab.2011.04.003. Epub 2011 May 5. English, French. PMID 21596642
- [Result] Bayen E, Pradat-Diehl P, Jourdan C, Ghout I, Bosserelle V, Azerad S, Weiss JJ, Joel ME, Aegerter P, Azouvi P; Steering Committee of the PariS-TBI study. Predictors of informal care burden 1 year after a severe traumatic brain injury: results from the PariS-TBI study. J Head Trauma Rehabil. 2013 Nov-Dec;28(6):408-18. doi: 10.1097/HTR.0b013e31825413cf. PMID 22691963
- [Result] Fugate LP, Spacek LA, Kresty LA, Levy CE, Johnson JC, Mysiw WJ. Measurement and treatment of agitation following traumatic brain injury: II. A survey of the Brain Injury Special Interest Group of the American Academy of Physical Medicine and Rehabilitation. Arch Phys Med Rehabil. 1997 Sep;78(9):924-8. doi: 10.1016/s0003-9993(97)90051-4. PMID 9305262
- [Result] Osiurak F, Jarry C, Allain P, Aubin G, Etcharry-Bouyx F, Richard I, Bernard I, Le Gall D. Unusual use of objects after unilateral brain damage: the technical reasoning model. Cortex. 2009 Jun;45(6):769-83. doi: 10.1016/j.cortex.2008.06.013. Epub 2008 Nov 8. PMID 19084221